CLINICAL TRIAL: NCT05020444
Title: A Phase I Clinical Trial With TriPRIL CAR T Cells for the Treatment of Patients With Relapsed or Refractory Multiple Myeloma
Brief Title: TriPRIL CAR T Cells in Multiple Myeloma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Marcela V. Maus, M.D.,Ph.D. (Other)
Responsible Party: Sponsor-Investigator, Marcela V. Maus, M.D.,Ph.D., Sponsor Investigator, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-518
Record Dates: First submitted 2021-08-18; First posted 2021-08-25 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Multiple Myeloma; Multiple Myeloma in Relapse; Refractory Multiple Myeloma
Keywords: Multiple Myeloma; Multiple Myeloma in Relapse; Refractory Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Cyclophosphamide; fludarabine; fludarabine phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TriPRIL CAR T Cells-Dose Escalation (Experimental): Prior to receiving TriPRIL CAR T Cells, participants will undergo two preparatory processes:
  * Leukapheresis: White blood cells will be collected and manufacture TriPRIL CAR T cells at a GMP manufacturing facility.
  * Lymphodepletion: On days, -5, -4. -3 participants will receive 3 days of chemotherapy to decrease the number of lymphocytes
  TriPRIL CAR T Cells will be administered intravenously on day 0 using a 3+3 dose escalation design
  Interventions: Drug: TriPRIL CAR T Cells; Drug: Cyclophosphamide; Drug: Fludarabine
- TriPRIL CAR T Cells-Dose Expansion (Experimental): Prior to receiving TriPRIL CAR T Cells, participants will undergo two preparatory processes:
  * Leukapheresis: White blood cells will be collected and manufacture TriPRIL CAR T cells at a GMP manufacturing facility.
  * Lymphodepletion: On days, -5, -4. -3 participants will receive 3 days of chemotherapy to decrease the number of lymphocytes
  TriPRIL CAR T Cells will be administered intravenously on day 0 using the respective dose (at or below the Maximum Tolerated Dose-MTD), as determined during the dose escalation part.
  Interventions: Drug: TriPRIL CAR T Cells; Drug: Cyclophosphamide; Drug: Fludarabine

INTERVENTIONS:
Drug: TriPRIL CAR T Cells — Intravenous infusion
Drug: Cyclophosphamide — Intravenous infusion
  Other Names: Cytoxan; Neosar
Drug: Fludarabine — Intravenous infusion
  Other Names: Fludara

SUMMARY:
This research study involves the study of TriPRIL CAR T Cells for treating people with relapsed or refractory multiple myeloma and to understand the side effects when treated with TriPRIL CAR T Cells.

This research study involves the study drugs:.

* TriPRIL CAR T Cells
* Fludarabine and Cyclophosphamide: Standardly used chemotherapy drugs as part of lymphodepleting process

DETAILED DESCRIPTION:
This is a two-part, non-randomized, open label, single-site Phase 1 study of TriPRIL CAR T Cells as a treatment for relapsed or refractory multiple myeloma.

This study consists of 2 parts:

* Part A (Dose Escalation) : The investigators are looking to find the highest dose of the study intervention that can be administered safely without severe or unmanageable side effects, not everyone who participates in this research study will receive the same dose of the study intervention. The dose given will depend on the number of participants who have been enrolled prior and how well the dose was tolerated Once determined, this highest dose will then be used in the dose expansion part of the study.
* Part B (Expansion Cohort):Participants will be treated at the respective dose as determined during Part A (Dose Escalation).

TriPRIL CAR T Cells is an investigational treatment that uses a person's own immune cells, called T cells, to try to kill their cancerous cells. T cells fight infections and can also kill cancer cells in some cases. The U.S. Food and Drug Administration (FDA) has not approved TriPRIL CAR T Cells as a treatment for any disease.This is the first time that TriPRIL CAR T Cells will be given to humans.

The research study procedures include screening for eligibility and study treatment including evaluations and follow up visits.

Participants will receive one infusion of the study treatment and will be followed for up to 2 years.

It is expected that about 18 people will take part in this research study.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and the willingness to sign a written informed consent document.
* Age ≥18 years at the time of signing informed consent.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Life expectancy of greater than 12 weeks
* Histologically or cytologically confirmed diagnosis of relapsed/refractory multiple myeloma. Documented measurable disease includes at least one or more of the following criteria:

  * Serum M-protein ≥1.0 g/dL
  * Urine M-protein ≥200 mg/24 hours
  * Involved serum free light chain ≥100 mg/L with abnormal κ/λ ratio
  * Bone marrow plasma cells ≥30%
* Relapsed/refractory multiple myeloma with at least 3 prior regimens of systemic therapy including proteasome inhibitor, IMiDs and anti-CD38 antibody; or has "triple-refractory" disease following treatment with proteasome inhibitor, IMiD and anti-CD38 antibody, as part of the same or different regimens.

Note: IMWG criteria defines refractory disease as disease progression on or within 60 days of receiving a therapy Note: Induction treatment with or without hematopoietic stem cell transplant and with or without maintenance is considered a single regimen.

* Adequate organ and marrow function as defined below:

  * O2 saturation ≥92% on room air while awake
  * LVEF ≥40% by ECHO or MUGA scan
  * ANC ≥1.0k/μl, PLT ≥50k/μl, (NOTE: Platelet transfusion not allowed within 7 days; growth factor neupogen not allowed within 7 days, neulasta within 14 days)
  * Creatinine clearance ≥30 mL/min and not on dialysis
  * AST/ALT <3 x ULN
  * Direct bilirubin <1.5 x ULN (allow x 3 ULN for Gilbert's syndrome)
  * PTT, PT/INR <1.5 x ULN, unless on a stable dose of anti-coagulant for a thromboembolic event (Patients with any history of thromboembolic stroke; or history or Grade 2 or greater hemorrhage within 60 days are excluded)
* Resolution of AEs from any prior therapy to ≤ Grade 1 (≤ G2 alopecia and ≤ G2 sensory neuropathy are allowed, cytopenias allowed per eligibility criteria above)
* Participants with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
* The effects of TriPRIL CAR T cells on the developing human fetus are unknown. Male and female participants of childbearing potential must agree to use highly effective methods of birth control prior to study entry, for the duration of study participation, and through 6 months after completion of TriPRIL CAR T cells administration. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.

NOTE: Highly effective contraception methods include:

* Total abstinence
* Female sterilization (tubal ligation, bilateral oophorectomy, and/or hysterectomy)
* Male sterilization, at least 6 months prior to screening
* Intrauterine device
* Oral, injected, or implanted hormonal contraception AND barrier methods of contraception

  * Willing to comply with and able to tolerate study procedures, including Long-term Safety Follow-up lasting up to 15 years per FDA guidance

Exclusion Criteria:

* Treatment with any of the following therapies as specified below:

  * Any prior systemic treatment for multiple myeloma within the 14 days prior to scheduled leukapheresis unless discussed with the medical monitor
  * Receiving high-dose (e.g., >10 mg prednisone or equivalent) systemic steroid therapy or any other form of immunosuppressive therapy within 14 days prior to leukapheresis
  * Autologous stem cell transplantation within 3 months prior to leukapheresis
  * Any prior allogeneic stem cell transplantation
  * Other CAR-T cell therapy within 6 months of leukapheresis
* Plasma cell leukemia or history of plasma cell leukemia
* Patients with extramedullary disease only without meeting criteria for measurable disease as per inclusion criteria above.
* No Bispecific T cell engagers withing 6 months of apheresis
* No bendamustine within 6 months of apheresis
* Patients with solitary plasmacytomas without evidence of other measurable disease
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to CAR- T cells
* Contraindication to the protocol-specified doses of fludarabine or cyclophosphamide
* Participants who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > Grade 1) with the exception of ≤ G2 alopecia and grade ≤2 sensory neuropathy.
* Active bacterial, viral, or fungal infection requiring systemic treatment (isolated fever may not constitute active infection in and of itself, e.g., related to disease)
* Symptomatic congestive heart failure
* Unstable angina, arrhythmia, or myocardial infarction (MI) within 6 months prior to screening
* Significant pulmonary dysfunction
* Auto-immune disease requiring immunosuppressive therapy
* Pulmonary embolism or DVT within three months of enrollment or uncontrolled thromboembolic events. Therapeutic dosing of anticoagulants (e.g., warfarin, low molecular weight heparin, Factor Xa inhibitors) is allowed for history of DVT or PE if greater than three months from time of enrollment. Prophylactic anticoagulation is allowed.
* Recent severe hemorrhage (within the past 60 days)
* Seropositive for and with evidence of active hepatitis B or C infection at time of screening, or HIV seropositive

  * Subjects with a history of hepatitis B but have received antiviral therapy and have non-detectable viral DNA for 6 months are eligible
  * Subjects seropositive because of hepatitis B virus vaccine with no signs or active infection are eligible
  * Subjects who had hepatitis C but have received antiviral therapy and show no detectable HCV viral RNA for 6 months are eligible
* Active central nervous system (CNS) involvement by malignancy. NOTE: subjects who are asymptomatic, stable, and received prior effective treatment for CNS disease may be eligible after discussion with the medical monitor.
* Any sign of active or prior CNS pathology including history of epilepsy, seizure, paresis, aphasia, stroke, subarachnoid hemorrhage or CNS bleed, severe brain injury, dementia, cerebellar disease, Parkinson's disease, organic brain syndrome or psychosis.
* Active malignancy not related to myeloma that has required therapy in the last 3 years or is not in complete remission. Exceptions to this criterion include successfully treated non-metastatic basal cell or squamous cell skin carcinoma, or prostate cancer that does not require therapy. Other similar malignant conditions may be discussed with and permitted by the medical monitor.
* Females who are pregnant or breastfeeding or females of childbearing potential not using an effective method of birth control
* Subjects with any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from participating in study (or full access to medical records) as written including follow up, the interpretation of data or place the subject at unacceptable risk
* Participants taking any other medicine concurrently that may interfere with the study (need to consult with the principle investigator)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2021-10-05 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | Week 24 post dosing, and every three months until two years.
  Study-related adverse events (AEs) will be listed and tabulated by type and study cohort. The rate of AEs in all infused patients, both within study cohorts and overall, will be calculated and reported with exact 95% confidence intervals. A separate safety analysis will report similar information within patients infused at the target dose of 1x108 or 3x108 TriPRIL CAR T cells.
Incidence of Dose Limiting Toxicity (DLT) | Week 24 post dosing, and every three months until two years.
  Dose-limiting toxicities will be listed and tabulated by type and study cohort.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | 1 month, 6 months, 12 months, and 24 after CAR T cell treatment.
  Data will be listed, tabulated, and presented descriptively using Kaplan Meier plots.
Overall Survival (OS) | 1 month, 6 months, 12 months and 24 months after CAR T cell treatment.
  Data will be listed, tabulated, and presented descriptively using Kaplan Meier plots.
Progression Free Survival (PFS) | 1 month, 6 months, 12 months and 24 months after CAR T cell treatment.
  Data will be listed, tabulated, and presented descriptively using Kaplan Meier plots.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J Frigault, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital Cancer Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation